CLINICAL TRIAL: NCT02313090
Title: Study of Welltang- a Cell Phone-based Diabetes Management Application's Effect on Blood Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhou Weibin, Prime investigator, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ChiCTR-IOR-14005515
Record Dates: First submitted 2014-11-25; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Welltang (Experimental): patients using Welltang
  Interventions: Other: Welltang
- usual standard care (No Intervention): patients under usual standard of diabetic care

INTERVENTIONS:
Other: Welltang — The intervention group installed Welltang (downloaded from www.welltang.com for free) designed by Shanghai Geping Information and Technique Company Ltd (Shanghai, China) on their cell phones. Welltang is a cell phone- based diabetes management application that consists of three main parts: knowledge, self-management, communication between patients and clinicians
  Arms: Welltang

SUMMARY:
The aim was to assess the impact of a cell phone-based diabetes management application (Welltang) on HbA1c, blood glucose, lipids, physical activity, weight, and blood pressure during 3 months. And hypoglycemic events, the satisfaction of the patients with Boyibang, their diabetes knowledge and self-care behaviors were also evaluated.

DETAILED DESCRIPTION:
At baseline, all patients completed the Diabetes Self- Care Behavior Questionnaire and a Diabetes Knowledge Survey. Health, medical and demographic history, height and weight, waist and hip circumferences, and blood pressure were recorded. HbA1c and low-density lipoprotein cholesterol (LDL-C) level were tested. All of these data were measured 3 months later at the conclusion of the study intervention.

ELIGIBILITY:
Inclusion Criteria:

* All diabetes, aged more than 18 years old. No limit for HbA1c was defined

Exclusion Criteria:

* patients have any severe complications such as end phase of diabetic nephropathy or proliferative retinopathy. patients who cannot use smart phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
blood pressure | 3 months
low density lipoprotein cholesterol | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Weibin Zhou, phD, Principal Investigator — the First Affiliated Hospital to Zhejiang University School of Medicine